CLINICAL TRIAL: NCT04804865
Title: Secondary Prognostic Index in RefrActory Diffuse Large B Cells Lymphoma
Brief Title: Secondary Prognostic Index in RefrActory Lymphoma
Acronym: SPiRAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Other Study IDs: WP-2019-02
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Diffuse Large B Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: prognostic score; cancer
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- population: The population includes adult patients.
  * Patients died from refractory or relapsed diffuse large-cell lymphoma.
  * Patients <65 years of age eligible for an autologous transplant should have relapsed after the autologous transplant.
  * Patients >65 years of age or not eligible after an autologous transplant must have received at least one RCHOP-type treatment line (2 cycles).
  Interventions: Other: prognostic assessment

INTERVENTIONS:
Other: prognostic assessment — determination of a prognostic score with 3 clinical and 5 biological parameters.

SUMMARY:
60% of patients with diffuse large B cell lymphoma are healed after first-line treatment which whatever the age. For the remaining 40% of patients (relapses and primary refractories):

* 38% of patients will be cured with a 2nd line including an autologous haematopoietic cell transplantation for those under 65 years.
* for older patients who are not eligible for a autograft: only 70% of patients will be able to receive 2nd line treatment with rates response less than 50%.
* the survival rate in patients receiving 3rd line treatment or more is 15% at 2 years. Actually, no standard of chemotherapy is offered to relapsed or refractory patients after 2 therapeutic lines. Subsequent lines lead to hospitalizations for infectious complications or transfusions without clear clinical benefit with often an impacted quality of life.

Palliative care is rarely offered as part of the treatment overall load.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* died of diffuse large B cell lymphoma
* Refractory or relapsing after 2 treatment lines for young patients (RCHOP then recovery with platinum salts and autograft) and one line for elderly patients (RCHOP)

Exclusion Criteria:

* patients with HIV infection
* solid tumor treated less than 5 years ago with the exception of skin carcinoma or carcinoma in situ of the uterine cervix treated locally
* inclusion in a therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes adult patients, who have died with refractory or relapsed diffuse large-cell lymphoma. Patients <65 years of age eligible for an autologous transplant should have relapsed after the autologous transplant.
  Patients> 65 years of age or not eligible after an autologous transplant must have received at least one RCHOP-type treatment line (2 cycles).
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Time between the date of relapse or no response observed (after 2 lines of chemotherapy in young patients and one line for elderly patients) and the date of death regardless of the cause.

SECONDARY OUTCOMES:
Median response time after each line | 5 years
  Time between the date when the first response criterion is observed (partial or complete response) and the date when the recurrence or progression is objectively documented
Event-free survival since diagnosis and after each line of treatment received | 5 years
  Time between the date of diagnosis and the date of the first event observed, then between the date of the first administration of each line of treatment administered and the date of onset of the first event observed.
the intensity dose of chemotherapy received | 6 month
  Total amount of chemotherapy administered relative to the theoretical dose calculated according to the patient's body surface area.
the Cumulative Illness Rating Scale for comorbidities score in patients over 65 years old | 6 month
  The cumulative illness rating scale for comorbidity score in elderly patients will be calculated according to the table proposed by Salvi et al. in 2008 (values :0 to 56; higher scores mean a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DU, MD, Study Director — Weprom
Locations (2):
- France (2):
  - Clinique Victor Hugo / Centre Jean Bernard, Le Mans
  - Centre d'Oncologie de Gentilly, Nancy

IPD SHARING:
Plan to Share IPD: No